CLINICAL TRIAL: NCT01819272
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Assess the Efficacy, Safety, and Tolerability of Delayed-Release Metformin in Subjects With Type 2 Diabetes Mellitus
Brief Title: Assessing the Efficacy, Safety, and Tolerability of Met DR in Subjects With T2DM Over 12 Weeks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elcelyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCRM105
Record Dates: First submitted 2013-03-19; First posted 2013-03-27 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 600 mg DR (Experimental): 600 mg delayed-release metformin once daily in the morning
  Interventions: Drug: Met DR
- 800 mg DR (Experimental): 800 mg delayed-release metformin once daily in the morning
  Interventions: Drug: Met DR
- 1000 mg DR (Experimental): 1000 mg delayed-release metformin once daily in the morning
  Interventions: Drug: Met DR
- 1000 mg XR (Active Comparator): 1000 mg extended-release metformin once daily in the evening
  Interventions: Drug: Met XR
- 2000 mg XR (Active Comparator): 2000 mg extended-release metformin once daily in the evening
  Interventions: Drug: Met XR
- Placebo (Placebo Comparator): Placebo once daily in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Met DR — metformin delayed-release tablets
  Arms: 1000 mg DR; 600 mg DR; 800 mg DR
Drug: Met XR — metformin extended-release tablets
  Arms: 1000 mg XR; 2000 mg XR
Drug: Placebo — placebo delayed-release tablets
  Arms: Placebo

SUMMARY:
This study compared the effect of delayed-release metformin (Met DR) to placebo and extended release metformin (Met XR) on glycemic control (fasting plasma glucose and HbA1c) and body weight, and assessed the safety and tolerability of a range of doses of Met DR when administered in subjects with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with T2DM who was ≥18 and ≤65 years of age at Visit 1
2. Had a body mass index (BMI) of 25.0 kg/m² to 45.0 kg/m², inclusive, at Visit 1
3. Screening HbA1c 7.0 to 9.5% (inclusive) at Visit 1 if treated with diet and exercise alone, or 6.0 to 9.5% (inclusive) if on a stable dose of either metformin or DPP-4 inhibitor monotherapy for a minimum of 2 months at Visit 1, or a combination of these 2 agents only on a stable regimen for a minimum of 2 months at Visit 1
4. Had serum creatinine concentration of <1.5 mg/dL (male) or <1.4 mg/dL (female) and an estimated glomerular filtration rate (eGFR) of ≥60 mL/min/1.73 m² based on the Modification of Diet in Renal Disease (MDRD) equation
5. Had a fasting glucose concentration of <280 mg/dL at Visit 1
6. Had a stable body weight, i.e., not varying by >5% for at least 6 months prior to Visit 1 as documented by the investigator
7. Was male, or if female and met all of the following criteria:

   1. Not breastfeeding
   2. Negative pregnancy test result (human chorionic gonadotropin, beta subunit [βhCG]) at Visit 1 (not applicable to hysterectomized females)
   3. If of child bearing potential (including perimenopausal women who have had a menstrual period within 1 year), must have practiced and be willing to continue to practice appropriate birth control during the entire duration of the study
8. Had a physical examination and ECG with no clinically significant abnormalities as judged by the investigator at Visit 1
9. Had no clinically significant laboratory test values (clinical chemistry, hematology, urinalysis) other than those expected in subjects with diabetes as judged by the investigator at Visit 1
10. Either was not treated with or had been on a stable treatment regimen with any of the following medications for a minimum of 2 months prior to Visit 1:

    1. Hormone replacement therapy (female subjects)
    2. Oral contraceptives (female subjects)
    3. Antihypertensive agents
    4. Lipid-lowering agents
    5. Thyroid replacement therapy
    6. Antidepressant agents
    7. Testosterone therapy (male subjects)
11. If on chronic thyroid pharmacologic therapy, had a serum thyroid-stimulating hormone test result within the normal range at Visit 1
12. Was willing and able to follow study procedures
13. Was able to read, understand, and sign the Informed Consent Form and an Authorization to Use and Disclose Protected Health Information form, answer the study questions, communicate with the investigator, and understand and comply with protocol requirements

Exclusion Criteria:

1. Had a clinically significant medical condition that could potentially affect study participation and/or personal well-being, as judged by the investigator, including but not limited to the following conditions:

   1. Hepatic disease
   2. Renal disease
   3. Gastrointestinal disease
   4. Endocrine disorder except T2DM
   5. Cardiovascular disease
   6. Central nervous system diseases
   7. Psychiatric or neurological disorders
   8. Organ transplantation
   9. Chronic or acute infection (e.g., tuberculosis, human immunodeficiency virus, hepatitis B virus, or hepatitis C virus)
   10. Orthostatic hypotension, fainting spells or blackouts
   11. Allergy or hypersensitivity
2. Clinically significant malignant disease (with the exception of basal and squamous cell carcinoma of the skin) within 5 years of Visit 1
3. Had known hypersensitivity, intolerability, or allergies to metformin HCl or any component of study treatment
4. Had a physical, psychological, or historical finding that, in the investigator's opinion, would make the subject unsuitable for the study
5. Current drugs or alcohol abuse or had a history of abuse that in the investigator's opinion would cause the individual to be noncompliant with study procedures
6. Had major surgery or a blood transfusion within 2 months of Visit 1 or was planning to donate blood during the study, or had a significant blood loss within 2 months prior to Visit 1
7. Had been treated, was being treated, or was expected to require or undergo treatment with any of the following excluded medications:

   1. Insulin or sulphonylurea treatment within 3 months of Visit 1
   2. GLP-1 receptor agonists and/or thiazolidinedione treatment within 6 months of Visit 1
   3. Nifedipine within 3 months of Visit 1
   4. Systemic corticosteroids by oral, intravenous, intra-articular, or intra-muscular route within 30 days of screening or for more than 1 week within 3 months of Visit 1
   5. Prescription weight loss medications within 3 months of Visit 1
   6. Chronic or frequent use, in the judgment of the investigator, of any drug treatment that affects gastric pH (prescription or over-the-counter), including proton pump inhibitors or any antacids or medications such as Rolaids or Pepcid within 1 month of Visit 1
   7. Had received or planned to receive any iodinated contrast dye within 1 week prior to Visit 1 (Screening)
8. Had a surgical gastrointestinal procedure that may impact the gut hormonal response to study medication
9. History or presence of inflammatory bowel disease or other severe gastrointestinal disease, particularly those which may impact gastric emptying, such as gastroparesis, pyloric stenosis, gastric bypass surgery or gastric banding surgery
10. Had received any investigational drug within 30 days (or five half-lives of the investigational drug, whichever was greater) of Visit 1
11. Was an immediate family member (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the clinical study site, or was directly affiliated with the study at the clinical study site
12. Was employed by Elcelyx Therapeutics, Inc. (that is an employee, temporary contract worker, or designee responsible for the conduct of the study)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lewin, Principal Investigator — National Research Institute - Wilshire; Rubin Saavedra, Principal Investigator — Alliance Against Diabetes / AAD Clinical Research; Lydie Hazan, Principal Investigator — Axis Clinical Trials; Robert Lipetz, Principal Investigator — Encompass Clinical Research; Audrey Lacour, Principal Investigator — Juno Research, LLC - Houston; Donald Hurley, Principal Investigator — Medical Research South, LLC; Eli M Roth, Principal Investigator — Sterling Research Group, Ltd. - Auburn; Robert Strzinek, Principal Investigator — Protenium Clinical Research, LLC; Richard Marple, Principal Investigator — Castlerock Clinical Research Consultants, LLC; Farah Sultan, Principal Investigator — Achieve Clinical Research, LLC; Thomas Moretto, Principal Investigator — American Health Network - Indianapolis; Azazuddin A Ahmed, Principal Investigator — Apex Medical Research - Illinois; Cynthia Strout, Principal Investigator — Coastal Carolina Research Center; John Pullman, Principal Investigator — Big Sky Clinical Research; Gregory Collins, Principal Investigator — Charlotte Clinical Research; David Hassman, Principal Investigator — Comprehensive Clinical Research; Leonard Zemel, Principal Investigator — Creekside Endocrine Associates; Diane Smith, Principal Investigator — CSRA Partners in Health, Inc.; Julio Rosenstock, Principal Investigator — Dallas Diabetes and Endocrine Center; David Johnson, Principal Investigator — Searcy Medical Center; Stephen Ong, Principal Investigator — MD Medical Research; Cynthia Huffman, Principal Investigator — Meridien Research - Tampa; Ramon Vargas, Principal Investigator — New Orleans Center for Clinical Research; Almena Free, Principal Investigator — Pinnacle Research Group; Douglas Short, Principal Investigator — PMG Research of Raleigh, LLC; Jonathan Wilson, Principal Investigator — PMG Research of Winston-Salem, LLC; Alexander White, Principal Investigator — Progressive Medical Research; Ronald Brazg, Principal Investigator — Rainier Clinical Research Center; Matthew Davis, Principal Investigator — Rochester Clinical Research; Charles Fogarty, Principal Investigator — Spartanburg Medical Research; Ralph DeFronzo, Principal Investigator — The University of Texas Health Science Center at San Antonio; Craig S Thompson, Principal Investigator — Craig S Thompson MD LLC; Subodh Bhuchar, Principal Investigator — Pioneer Research Solutions Inc.; Susan Greco, Principal Investigator — Jacksonville Center For Clinical Research; Harold Bays, Principal Investigator — Louisville Metabolic and Atherosclerosis Research Center; Barry Lubin, Principal Investigator — National Clinical Research - Norfolk, Inc.; Mark Christiansen, Principal Investigator — Diablo Clinical Research, Inc.; Andrea Lawless, Principal Investigator — Biofortis, Inc.; Kathryn J Lucas, Principal Investigator — Diabetes and Endocrinology Consultants, P.C.; Hugo Toro, Principal Investigator — Juno Research, LLC - Katy; Eva M Heurich, Principal Investigator — Compass Research, LLC; Chander Arora, Principal Investigator — RAS Health Ltd; Patricia Buchanan, Principal Investigator — Willamette Valley Clinical Studies; Thomas Blevins, Principal Investigator — Texas Diabetes & Endocrinology, P.A. - Austin; Anna Chang, Principal Investigator — John Muir Physician Network Clinical Research Center; John Hoekstra, Principal Investigator — National Clinical Research - Richmond, Inc.; Lyle Myers, Principal Investigator — Kentucky Diabetes Endocrinology Center; Stephanie Shaw, Principal Investigator — Texas Diabetes and Endocrinology, P.A. - Round Rock; Purvi Mehra, Principal Investigator — eStudySite; Traci Turner, Principal Investigator — Metabolic and Atherosclerosis Research Center

REFERENCES:
- [Background] Buse JB, DeFronzo RA, Rosenstock J, Kim T, Burns C, Skare S, Baron A, Fineman M. The Primary Glucose-Lowering Effect of Metformin Resides in the Gut, Not the Circulation: Results From Short-term Pharmacokinetic and 12-Week Dose-Ranging Studies. Diabetes Care. 2016 Feb;39(2):198-205. doi: 10.2337/dc15-0488. Epub 2015 Aug 18. PMID 26285584

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 600 mg DR | 800 mg DR | 1000 mg DR | 1000 mg XR | 2000 mg XR
Started | 41 | 39 | 40 | 40 | 40 | 40
Completed | 35 | 36 | 37 | 35 | 36 | 33
Not Completed | 6 | 3 | 3 | 5 | 4 | 7
Not completed — Adverse Event | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 1 | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 2 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 0 | 1 | 2 | 1 | 0 | 1
Not completed — Loss of Glucose Control | 2 | 1 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 600 mg DR | 800 mg DR | 1000 mg DR | 1000 mg XR | 2000 mg XR | Total
Number analyzed (Participants) | 41 | 39 | 40 | 40 | 40 | 40 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (10.22) | 53.5 (8.34) | 52.6 (9.69) | 51.8 (9.05) | 51.0 (9.62) | 52.0 (9.53) | 52.0 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 27 | 14 | 22 | 21 | 127
  Male | 19 | 18 | 13 | 26 | 18 | 19 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 10 | 14 | 10 | 10 | 75
  Not Hispanic or Latino | 24 | 25 | 30 | 26 | 30 | 30 | 165
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 3 | 0 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 11 | 9 | 13 | 9 | 14 | 12 | 68
  White | 28 | 30 | 23 | 30 | 24 | 27 | 162
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 2
BMI [Mean (Standard Deviation); unit: kg/m²] | 33.6 (5.28) | 33.1 (5.74) | 33.5 (5.86) | 33.3 (5.55) | 32.8 (5.27) | 33.7 (5.22) | 33.3 (5.44)
Previous T2DM Regimen [Number; unit: participants]
  Diet and exercise alone | 3 | 7 | 2 | 4 | 6 | 5 | 27
  DPP-4 inhibitor alone | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Metformin alone | 35 | 29 | 35 | 36 | 30 | 33 | 198
  Metformin/DPP-4 inhibitor combination | 3 | 2 | 3 | 0 | 4 | 2 | 14
Screening Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 146.5 (36.70) | 147.5 (42.56) | 142.4 (34.60) | 141.4 (29.79) | 139.0 (34.22) | 148.9 (41.36) | 144.3 (36.57)
Screening HbA1c [Mean (Standard Deviation); unit: %] | 7.19 (0.838) | 7.27 (0.864) | 7.17 (0.829) | 7.13 (0.899) | 7.10 (0.819) | 7.17 (0.869) | 7.17 (0.846)
Baseline Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 176.5 (54.70) | 180.1 (49.72) | 162.9 (40.10) | 172.3 (44.45) | 165.7 (50.01) | 180.3 (57.52) | 173.0 (49.72)
Baseline HbA1c [Mean (Standard Deviation); unit: %] | 7.40 (0.951) | 7.45 (0.887) | 7.33 (0.908) | 7.37 (0.890) | 7.36 (0.997) | 7.38 (0.980) | 7.38 (0.928)

OUTCOME MEASURES:

1. Primary Outcome: Change in Fasting Plasma Glucose (mg/dL) at 4 Weeks
Time Frame: Baseline and 4 weeks after the first dose of study medication
Population: Week 4 Evaluable
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | 600 mg DR | 800 mg DR | 1000 mg DR | 1000 mg XR | 2000 mg XR
Number analyzed (Participants) | 37 | 35 | 37 | 36 | 35 | 35
mg/dL | -4 [-69 to 48] | -11 [-124 to 150] | -13 [-62 to 145] | -18 [-90 to 113] | -12 [-111 to 58] | -25 [-110 to 20]
Statistical Analysis 1: Comparison: Placebo vs 600 mg DR; Test type: Superiority or Other; p = 0.0670, Kruskal-Wallis — p-value for pair-wise comparison without adjustment; Hodges-Lehmann Estimation = -9.0, 95% CI 2-sided [-21.0 to 1.0]
Statistical Analysis 2: Comparison: Placebo vs 800 mg DR; Test type: Superiority or Other; p = 0.0057, Kruskal-Wallis — p-value for pair-wise comparison without adjustment; Hodges-Lehmann Estimation = -14.0, 95% CI 2-sided [-22.0 to -4.0]
Statistical Analysis 3: Comparison: Placebo vs 1000 mg DR; Test type: Superiority or Other; p = 0.1095, Kruskal-Wallis — p-value for pair-wise comparison without adjustment; Hodges-Lehmann Estimation = -12.0, 95% CI 2-sided [-25.0 to 3.0]
Statistical Analysis 4: Comparison: Placebo vs 1000 mg XR; Test type: Superiority or Other; p = 0.0097, Kruskal-Wallis — p-value for pair-wise comparison without adjustment; Hodges-Lehmann Estimation = -12.0, 95% CI 2-sided [-23.0 to -3.0]
Statistical Analysis 5: Comparison: Placebo vs 2000 mg XR; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis — p-value for pair-wise comparison without adjustment; Hodges-Lehmann Estimation = -28.0, 95% CI 2-sided [-42.0 to -17.0]

2. Secondary Outcome: AUC4-12wk of Change in Fasting Plasma Glucose (mg/dL*Week) Concentrations From Baseline to 12 Weeks
Time Frame: Baseline and 4 to 12 weeks after the first dose of study medication
Population: Week 12 Evaluable
Measure: Median (Full Range); unit: mg/dL*week
Arm/Group | Placebo | 600 mg DR | 800 mg DR | 1000 mg DR | 1000 mg XR | 2000 mg XR
Number analyzed (Participants) | 30 | 34 | 37 | 34 | 31 | 30
mg/dL*week | 4.00 [-784.0 to 698.0] | -96.00 [-894.0 to 414.0] | -108.00 [-556.0 to 612.0] | -156.00 [-782.0 to 522.0] | -98.00 [-880.0 to 314.0] | -215.00 [-856.0 to 186.0]
Statistical Analysis 1: Comparison: Placebo vs 600 mg DR; Test type: Superiority or Other; p = 0.0226, Kruskal-Wallis — p-value for pair-wise comparison without adjustment; Hodges-Lehmann Estimation = -106.0, 95% CI 2-sided [-208.0 to -16.00]
Statistical Analysis 2: Comparison: Placebo vs 800 mg DR; Test type: Superiority or Other; p = 0.0068, Kruskal-Wallis — p-value for pair-wise comparison without adjustment; Hodges-Lehmann Estimation = -106.0, 95% CI 2-sided [-180.0 to -32.00]
Statistical Analysis 3: Comparison: Placebo vs 1000 mg DR; Test type: Superiority or Other; p = 0.0071, Kruskal-Wallis — p-value for pair-wise comparison without adjustment; Hodges-Lehmann Estimation = -152.0, 95% CI 2-sided [-252.0 to -42.00]
Statistical Analysis 4: Comparison: Placebo vs 1000 mg XR; Test type: Superiority or Other; p = 0.0405, Kruskal-Wallis — p-value for pair-wise comparison without adjustment; Hodges-Lehmann Estimation = -101.0, 95% CI 2-sided [-208.0 to -4.00]
Statistical Analysis 5: Comparison: Placebo vs 2000 mg XR; Test type: Superiority or Other; p < .0001, Kruskal-Wallis — p-value for pair-wise comparison without adjustment; Hodges-Lehmann Estimation = -224.0, 95% CI 2-sided [-334.0 to -118.0]

3. Secondary Outcome: Change in HbA1c (%) at 12 Weeks
Time Frame: Baseline and 12 weeks after the first dose of study medication
Population: Week 12 Evaluable
Measure: Least Squares Mean (Standard Error); unit: HbA1c (%)
Arm/Group | Placebo | 600 mg DR | 800 mg DR | 1000 mg DR | 1000 mg XR | 2000 mg XR
Number analyzed (Participants) | 30 | 34 | 37 | 34 | 31 | 30
HbA1c (%) | 0.45 (0.137) | -0.03 (0.125) | 0.00 (0.121) | 0.10 (0.124) | 0.00 (0.132) | -0.21 (0.133)
Statistical Analysis 1: Comparison: Placebo vs 600 mg DR; Test type: Superiority or Other; p = 0.0100, ANCOVA; Factor for treatment and baseline HbA1c as a covariate; LS Mean = -0.48, 95% CI 2-sided [-0.85 to -0.12]
Statistical Analysis 2: Comparison: Placebo vs 800 mg DR; Test type: Superiority or Other; p = 0.0153, ANCOVA; Factor for treatment and baseline HbA1c as a covariate; LS Mean = -0.45, 95% CI 2-sided [-0.81 to -0.09]
Statistical Analysis 3: Comparison: Placebo vs 1000 mg DR; Test type: Superiority or Other; p = 0.0611, ANCOVA; Factor for treatment and baseline HbA1c as a covariate; LS Mean = -0.35, 95% CI 2-sided [-0.71 to 0.02]
Statistical Analysis 4: Comparison: Placebo vs 1000 mg XR; Test type: Superiority or Other; p = 0.0188, ANCOVA; Factor for treatment and baseline HbA1c as acovariate; LS Mean = -0.45, 95% CI 2-sided [-0.83 to -0.08]
Statistical Analysis 5: Comparison: Placebo vs 2000 mg XR; Test type: Superiority or Other; p = 0.0006, ANCOVA; Factor for treatment and baseline HbA1c as a covariate; LS Mean = -0.67, 95% CI 2-sided [-1.04 to -0.29]

ADVERSE EVENTS:
Time Frame: Approximately 83 to 107 days depending on the number of intervening days between study visits
Arm/Group | Placebo | 600 mg DR | 800 mg DR | 1000 mg DR | 1000 mg XR | 2000 mg XR
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/39 | 0/40 | 2/40 | 1/40 | 0/40
Other Adverse Events (participants affected / at risk) | 9/41 | 9/39 | 11/40 | 9/40 | 8/40 | 8/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | 600 mg DR (N=39) | 800 mg DR (N=40) | 1000 mg DR (N=40) | 1000 mg XR (N=40) | 2000 mg XR (N=40)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Intravascular haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | 600 mg DR (N=39) | 800 mg DR (N=40) | 1000 mg DR (N=40) | 1000 mg XR (N=40) | 2000 mg XR (N=40)
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 5 | 2 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 2 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 1 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2
rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study may be published by INSTITUTE, however the publication shall not disclose any SPONSOR Confidential Information, the INSTITUTE shall send the SPONSOR a copy of any such proposed publication 90 days prior to submission for publication, the INSTITUTE, on request of the SPONSOR, shall delete any SPONSOR Confidential Information in the proposed publication, and the INSTITUTE shall, on the SPONSOR's request, delay submission while the SPONSOR files applications for patents.